CLINICAL TRIAL: NCT04374279
Title: A Phase II Trial to Promote Recovery From COVID-19 With Endocrine Therapy
Brief Title: Trial to Promote Recovery From COVID-19 With Endocrine Therapy
Acronym: RECOVER
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited resources.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COV2003; IRB00249425 (Other: JHM IRB)
Record Dates: First submitted 2020-05-04; First posted 2020-05-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: COVID-19; SARS-CoV 2
Keywords: COVID-19; Coronavirus; COVID; SARS-COV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — bicalutamide

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to bicalutamide with standard of care, or standard of care alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of care and bicalutamide (Active Comparator): Randomized participants receive bicalutamide 150mg oral for 7 days, plus standard of care
  Interventions: Drug: Bicalutamide 150 Mg Oral Tablet
- Standard of care only (No Intervention): Randomized participants receive standard of care only.

INTERVENTIONS:
Drug: Bicalutamide 150 Mg Oral Tablet — Bicalutamide 150 mg by mouth daily for 7 days
  Other Names: Casodex
  Arms: Standard of care and bicalutamide

SUMMARY:
Patients with COVID-19 requiring inpatient hospitalization will be randomized to treatment with standard of care or standard of care + bicalutamide. This will be a randomized, open-label study to determine if bicalutamide improves the rate of clinical improvement in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* COVID-19 infection, confirmed by polymerase chain reaction (PCR) test <=3 days from enrollment
* Require inpatient hospitalization due to COVID-19 with minimal respiratory symptoms
* Able to provide informed consent

Exclusion Criteria:

* Unable to take oral medication
* Pregnant or breastfeeding
* On non-invasive positive pressure ventilation or mechanical ventilation at time of study entry
* Requiring ≥6L oxygen or respiratory rate ≥30
* Taking bicalutamide, any systemic hormonal therapy, or prophylactic treatment for COVID-19 within one month of study entry
* Known hypersensitivity to bicalutamide or its components.
* A past medical history of cirrhosis or AST/ALT/Alk phos/bilirubin > 3x the upper limit of normal
* Patients with a clinical history of myocardial infarction or congestive heart failure within 6 months, or with prior echocardiogram showing ejection fraction < 40%
* Patients currently on coumadin anticoagulants due to the potential for drug-drug interactions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who have clinical improvement at day 7 after randomization | up to 7 days
  Percentage of participants who are discharged from the hospital or if they have had at least a 2-point improvement on the World Health Organization (WHO) Ordinal Scale for Clinical Improvement. The WHO clinical improvement scale has a score range of 0-8 where, 0= uninfected, 1= ambulatory with no limitation of activities; 2= ambulatory with limitations to activities; 3= hospitalized, mild disease, with no oxygen therapy; 4= hospitalized, mild disease, with oxygen by mask or nasal prongs; 5= hospitalized, severe disease, with non-invasive ventilation or high-flow oxygen; 6= hospitalized, severe disease, with intubation and mechanical ventilation; 7= hospitalized, severe disease, with ventilation and additional organ support (pressors, dialysis, ECMO); 8= death

SECONDARY OUTCOMES:
All-cause mortality | 28 days
  Number of participants deceased for any cause
Duration of hospitalization | up to 60 days
  Number of calendar days in the hospital
Percentage of patients needing upgrade to the intermediate care unit (IMC) | up to 60 days
Duration of IMC stay | up to 60 days
  Number of calendar days in IMC
Percentage of patients needing upgrade to the intensive care unit (ICU) | up to 60 days
Duration of ICU stay | up to 60 days
  Number of calendar days in ICU
Number of participants requiring mechanical ventilation | up to 60 days
Duration of mechanical ventilation | up to 60 days
  Number of calendar days requiring mechanical ventilation
Number of participants experiencing adverse events | up to 60 days
  Number of participants who are COVID-19 positive, experiencing adverse events as defined by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Catherine H Marshall, MD/MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No